CLINICAL TRIAL: NCT04000633
Title: Nebulized Lidocaine Versus Placebo to Prevent Cough at Emergence From Anesthesia: a Double Blind Prospective Randomised Trial
Brief Title: Nebulized Lidocaine to Prevent Cough at Emergence From Anesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mongi Slim Hospital (Other)
Responsible Party: Principal Investigator, Mhamed Sami Mebazaa, professor, Mongi Slim Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: lidocaïne cough prevention
Record Dates: First submitted 2019-06-26; First posted 2019-06-27 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Cough, General Anesthesia, Extubation, Lidocaine, Sore Throat
MeSH Terms: conditions — Cough; Pharyngitis | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: 2 groups comparaison between nebulized lidocaine versus placebo for prevention of cough at emergence from general anesthesia and post extubation sore throat
Who Masked: Participant, Care Provider
Masking Description: The investigator will provide to the anesthesiologist 1 seringue containing either lidocaine or normal saline to be nebulized before induction of general anesthesia
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lidocaine group (Active Comparator): the patients of this group will recieve nebulization of 5 ml of 2% lidocaine prior to induction of general anesthesia
  Interventions: Drug: Lidocaine 2%
- Placebo group (Placebo Comparator): the patients of this group will recieve nebulization of 5 ml of normal saline prior to induction of general anesthesia
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Lidocaine 2% — the patients of this group will recieve nebulization of 5 ml of 2% lidocaine prior to induction of general anesthesia
  Arms: lidocaine group
Drug: Normal saline — Normal saline
  Arms: Placebo group

SUMMARY:
our study aimed to evaluate the effect of nebulized lidocaine to decrease the incidence of cough and sore throat after extubation after surgeries requiring endotracheal intubation.

DETAILED DESCRIPTION:
our study aimed to evaluate the effect of nebulized lidocaine to decrease the incidence of cough and sore throat after extubation after surgeries requiring endotracheal intubation.

This randomized controlled study will compare the effect of Lidocaine and placebo nebulization in the immediate pre operative period in order to evaluate the effectiveness in reducing post extubation cough and sore throat.

ELIGIBILITY:
Inclusion Criteria:

* age>18 years
* ASA status I or II

Exclusion Criteria:

* Unexpected difficult laryngoscopy
* Surgery>3 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
incidence of cough at emergence from general anesthesia | 30 minutes after the end of surgery
  evaluation of incidence of cough at emergence from general anesthesia

SECONDARY OUTCOMES:
incidence of sore throat | 24 hours after tracheal extubation
  evaluation of incidence of sore throat

CONTACTS AND LOCATIONS:
Overall Officials: Mhamed Sami Mebazaa, Professor, Principal Investigator — Mongi Slim Hospital
Locations (1):
- Mongi Slim Hospital, La Marsa, Tunis Governorate, Tunisia

IPD SHARING:
Plan to Share IPD: No